CLINICAL TRIAL: NCT03016208
Title: The Misoprostol Vaginal Insert Used in Standard Compared With Adjusted Criteria for Labour Induction in Term Pregnancies: a Non-interventional Case Control Study
Brief Title: The Misoprostol Vaginal Insert for Labour Induction
Status: Completed | Type: Observational
Sponsor: Asklepios Kliniken Hamburg GmbH (Other)
Responsible Party: Principal Investigator, Peter Schwaerzler, Principal investigator, Asklepios Kliniken Hamburg GmbH
Other Study IDs: Miso2017
Record Dates: First submitted 2017-01-08; First posted 2017-01-10 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Labour Induction

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Misoprostol vaginal insert for max. 24hrs: 69 patients matching the inclusion criteria and received MVI for labour induction for a maximum of 24 hours
  Interventions: Drug: Misoprostol vaginal insert
- Misoprostol vaginal insert for max. 10hrs: 69 patients matching the inclusion criteria and received MVI for labour induction for a maximum of 10 hours
  Interventions: Drug: Misoprostol vaginal insert

INTERVENTIONS:
Drug: Misoprostol vaginal insert

SUMMARY:
Objective: To compare the efficacy and safety of the misoprostol vaginal insert (MVI) for labour induction using standard (MVI-24) and adjusted (MVI-10) criteria.

Design: Non-interventional observational case control study.

Setting: Tertiary-care academic centre in Germany.

Population: A cohort of 138 pregnant women ≥ 37/0 weeks undergoing labour induction.

Methods: Induction of labour with MVI in a consecutive series of women using standard (MVI-24, n = 69) or adjusted (MVI-10, n = 69) criteria.

Main outcome measures: The primary outcomes were the time from induction to delivery and the caesarean section rate. The secondary outcomes included the need for additional measures to induce labour, uterine tachysystole, tocolysis, fetal scalp blood testing, meconium-stained amniotic fluid, umbilical arterial pH, and Apgar score.

ELIGIBILITY:
Inclusion Criteria:

* gynecologist's indication for induction
* informed consent
* ≥ 37 weeks of gestation
* singleton pregnancies
* cephalic presentation
* cervical Bishop score of < 5 before priming reassuring fetal heart rate

Exclusion Criteria:

* known hypersensitivity to prostaglandins
* uterine scar
* parity > 5
* any contraindication for vaginal delivery
* cephalopelvic disproportion
* placenta praevia
* chorioamnionitis
* antepartum bleeding of unknown etiology
* cardiopulmonary, renal, hepatic maternal disease
* glaucoma
* fetal congenital abnormalities

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A cohort of 138 pregnant women ≥ 37/0 weeks undergoing labour induction.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Time from induction to delivery in minutes | August 2016
Rate of participants receiving a caesarean section compared to all participants being induced | August 2016

SECONDARY OUTCOMES:
Number of participants with treatment-related tachysystole as assessed by cardiotocography | August 2016
Number of participants with treatment-related adverse events following tocolysis with Partusisten | August 2016
Number of participants with fetal compromise assessed by the APGAR-Score and the postpartum fetal pH-value | August 2016

IPD SHARING:
Plan to Share IPD: No